CLINICAL TRIAL: NCT02215135
Title: Corifollitropin Alfa in Combination With Elective Cryopreservation of All Embryos After GnRH Agonist Triggering of Final Oocyte Maturation in PCOS Patients- a Prospective, Observational Proof-of -Concept Study
Brief Title: Corifollitropin Alfa Application in PCOS Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKH-8302-101-DR-15
Record Dates: First submitted 2014-06-04; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: In Vitro Fertilization
Keywords: Corifollitropin alfa; polycystic ovarian syndrome (PCOS); controlled ovarian hyperstimulation (COS); GnRH antagonist protocol; Ovarian hyperstimulation syndrome (OHSS)
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Corifollitropin in PCOS (Experimental): In GnRH antagonist protocol, a single dose corifollitropin alfa was administered for ovarian stimulation following rFSH daily injection to stimulate follicle development. GnRH agonist was given to trigger final oocyte maturation when three follicles reached 17 mm in size. The IVF or ICSI was planned then all embryos were elective cryopreserved.
  Interventions: Drug: Corifollitropin alfa

INTERVENTIONS:
Drug: Corifollitropin alfa — In GnRH antagonist protocol, ovarian stimulation with single dose of 100μg (BW≦60 kg) or 150μg (BW> 60 kg) corifollitropin alfa (Elonva, SC), followed 1 week later (stimulation day 8) by a daily dose of rFSH to the day of GnRH agonist triggering final oocyte maturation.
  Other Names: elonva

SUMMARY:
Corifollitropin alfa, single dose administered sustains multiple follicular development for 7 days. However, It may induce ovarian hyperstimulation syndrome (OHSS), especially in high responder women such as patients of polycystic ovary syndrome (PCOS). In GnRH antagonist protocol with agonist triggering of final oocyte maturation, following embryo cryopreservation can almost eliminate the risk of OHSS. To decrease the injection burden and prevent OHSS in PCOS patients undergoing IVF treatment, ovarian hyperstimulation with Corifollitropin alfa in GnRH antagonist protocol and GnRH agonist triggering of final oocyte maturation, following elective embryo cryopreservation was designed in this study. The purpose of this trial was conducted to confirmed whether this novel protocol could prevent OHSS, decreased the injection burden of PCOS patients and single dose corifollitropin alfa could support multiple follicular growth for 7 days.

DETAILED DESCRIPTION:
BACKGROUNG: Ovarian hyperstimulation syndrome (OHSS) is the most serious complication of ovulation induction. Therefore, Corifollitropin alfa, long acting recombinant follicular stimulation hormone (rFSH) application in PCOS women is warning. However, corifollitropin alfa could decrease the injection burden of patients undergoing IVF/ICSI treatment. In previous studies, embryo cryopreservation following GnRH agonist triggering final oocyte maturation in GnRH antagonist protocol can almost eliminate the risk of OHSS. This study was designed to analyze whether ovarian hyperstimulation in PCOS women with Corifollitropin alfa in GnRH antagonist protocol and GnRH agonist triggering, following freezing all embryos can decrease the injection burden without OHSS complication.

PURPOSE: To assess whether single dose Corifollitropin alfa sustains multiple follicular growth for seven days in GnRH antagonist protocol application in PCOS women, following embryo cryopreservation after GnRH agonist triggering can decrease injection benefit without OHSS complication.

METHODS: This prospective ,single center, observational study, thirty to fifty PCOS women aged 20-38 years old, In GnRH antagonist protocol, a single dose corifollitropin alfa was administered for ovarian stimulation (S1, stimulation D1). Seven days later, rFSH was daily injected to stimulate follicle development according to the ovarian response. GnRH antagonist was administered daily from S5 until the day of final oocyte maturation. GnRH agonist was given to replace hCG to trigger final oocyte maturation when three follicles reached 17 mm in size. The IVF or ICSI was planned then all embryos were elective cryopreservation. Transfer of embryos was performed in a subsequent frozen-thawed ET cycles. Primary outcome measure was the incidence of OHSS. The secondary outcome measures were numbers of oocytes retrieval, numbers of embryos frozen and pregnancy rate of subsequent FET cycles.

ANTICIPATED RESULTS: Decreasing the injection burden and maximal oocytes were retrieved without severe OHSS complication.

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of PCOS was according Rotterdam criteria ( twoi of three) included:

* chronic anovulation manifested by the symptoms of oligomenorrhoea
* ultrasonographic evidence of polycystic enlarged ovary with over 10 peripherally located follicles of 3-8mm diameter around a dense central stroma
* hyperandrogenaemia (serum testosterone concentrations over 0.8 ng/ml) or clinical hyperandrogenism.

Exclusion Criteria:

* A diagnosis of congenital adrenal hyperplasia, Cushing's syndrome, androgen-producing tumours, hyperprolactinaemia and thyroid dysfunction were all excluded.
* patients older than 38 years or with serum FSH level over 12 mIU/ml.
* patients wiht previous ovarian surgery
* husband with non-obstructive azoospermia

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with severe OHSS | one month
  The patients were assessed for signs and symptoms of OHSS on 3, 6, and 9 days after oocyte retrieval including history taking, physical examination, ultrasound scan, and blood tests for hematocrit, complete blood counts.The severity of OHSS was according to the classification of Golan et al. [Golan A, Ron-el R, Herman A, Soffer Y, Weinraub Z, Caspi E.Ovarian hyperstimulation syndrome: an update review. ObstetGynecol Surv. 1989;44:430-40].

SECONDARY OUTCOMES:
numbers of oocytes retrieved | one month
embryo quality | one month
  Grade 1 embryos consisted of symmetrical blastomeres of approximately equal size and without anucleate fragments.
  Grade 2 embryos had blastomeres of even or uneven size and had 10% of the volume of embryos filled with anucleate fragments.
  Grade 3 embryos had anucleate fragments occupying between 10 and 50% of the volume of the embryos.
  Grade 4 embryos had anucleate fragments .50% of the volume of the embryos.
No. of embryo frozen | one month

OTHER OUTCOMES:
Clinical pregnancy rate in the frozen-thawed embryo transfer cycle | 6 months
  Serum β-HCG level was measured 14 days after embryo transfer. Clinical pregnancy was defined as the presence of fetal cardiac activity on transvaginal ultrasonography at 7 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiann-Loung Hwang, MD, Study Chair — Department of Obstetrics and Gynecology, Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Shin-Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan